CLINICAL TRIAL: NCT02431468
Title: A Randomized, Double-Blind,Placebo-Controlled, Phase 2 Study Assessing the Safety, Tolerability and Efficacy of Bryostatin in the Treatment of Moderately Severe to Severe Alzheimer's Disease
Brief Title: A Study Assessing Bryostatin in the Treatment of Moderately Severe to Severe Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotrope Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTRP-101-202
Record Dates: First submitted 2015-04-22; First posted 2015-05-01 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — bryostatin 1; Bryostatins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bryostatin 1 20ug (Experimental): Bryostatin 20 micrograms administered IV over 45 minutes every other week after 2 initial loading doses of 24 micrograms administered weekly. A total of 7 doses administered over 12 weeks.
  Interventions: Drug: Bryostatin 1
- Bryostatin 1 40ug (Experimental): Bryostatin 40 micrograms administered IV over 45 minutes every other week after 2 initial loading doses of 48 micrograms administered weekly. A total of 7 doses administered over 12 weeks.
  Interventions: Drug: Bryostatin 1
- Placebo (Placebo Comparator): Placebo administered IV over 45 minutes every other week after 2 initial doses administered weekly. A total of 7 doses administered over 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bryostatin 1 — The investigational drug product, bryostatin, is a sterile, pyrogen-free, lyophilized powder intended for IV infusion upon reconstitution and dilution. Placebo is a sterile, pyrogen-free, lyophilized powder intended for IV infusion upon reconstitution and dilution.
  Other Names: bryostatin
  Arms: Bryostatin 1 20ug; Bryostatin 1 40ug
Other: Placebo — The placebo is a sterile, pyrogen-free, lyophilized powder identical in appearance to the active drug, intended for IV infusion upon reconstitution and dilution.
  Arms: Placebo

SUMMARY:
This is a randomized double-blind placebo-controlled study comparing different doses of bryostatin for the treatment of moderately severe to severe Alzheimer's disease. The study is 15 weeks in duration, including a safety and efficacy evaluation 30 days after the last dose of study drug.

DETAILED DESCRIPTION:
This study will enroll 150 moderately severe to severe Alzheimer's disease subjects. Subjects will be randomly assigned 1:1:1 to treatment with two different doses of bryostatin 1 or placebo. The primary analysis will take place after 12 weeks of treatment (7 doses).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from caregiver and subject (if possible) or legally acceptable representative if different from caregiver
* Male and female subjects 55-85 years of age inclusive
* Cognitive deficit present for at least 2 years that meet the diagnostic criteria for probable Alzheimer's
* Mini Mental State Exam (MMSE-2) score of 4-15
* Patients must be able to perform at least one item on the Severe Impairment Battery Scale
* Neuroimaging (computerized tomography (CT) or Magnetic Resonance Imaging (MRI)) within the last 24 months consistent with a diagnosis of probable Alzheimer's disease (AD)
* Reliable caregiver(s) or informant(s) who attends the subject at least an average of 3 hours or more per day for 3 or more days per week
* Adequate vision and motor function to comply with testing
* If taking drugs approved for treatment of Alzheimer's disease (e.g. cholinesterase inhibitors, memantine), must be on a stable dose for at least 3 months prior to entry into study and the dose must not change during the study unless a change is required due to an adverse event or a clinically significant change in the patient's status.

Exclusion Criteria:

* Dementia due to any condition other than AD, including vascular dementia (Rosen-modified Hachinski lschemic score ≥ 5)
* Evidence of significant central nervous system (CNS) vascular disease on previous neuroimaging including but not limited to: cortical stroke, multiple infarcts, localized single infarcts in the thalamus, angular gyrus, multiple lacunar infarcts or extensive white matter injury
* Clinically significant neurologic disease or condition other than AD, such as cerebral tumor, chronic subdural fluid collections, Huntington's Disease, Parkinson's Disease, normal pressure hydrocephalus, or any other diagnosis that could interfere with assessment of safety and efficacy
* Evidence of clinically significant unstable cardiovascular, pulmonary, renal, hepatic, gastrointestinal, neurologic, or metabolic disease within the 6 months prior to enrollment
* Poorly controlled diabetes, at the discretion of the Principal Investigator
* Creatinine clearance (CL) of <45ml/min
* Use of an active Alzheimer's vaccine within 2 years prior to screening
* Use of a monoclonal antibody for treatment of AD within 1 year prior to screening
* Any medical or psychiatric condition that is likely to require initiation of additional medication or surgical intervention during the course of the study
* Use of an investigational drug within 30 days prior to screening
* Prior exposure to bryostatin, or known sensitivity to bryostatin or any ingredient in the study drug
* Any other concurrent medical condition, which in the opinion of the PI makes the subject unsuitable for the clinical study

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Xenoscience, Inc/ 21st Century Neurology, Phoenix, Arizona
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Nader Pharmacology Research Institute, Los Alamitos, California
  - San Francisco Clinical Research Center, San Francisco, California
  - JEM Research, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of South Florida, Fort Myers, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Miami Jewish Health System, Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Compass Research, LLC, Orlando, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Compass Research, The Villages, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Alexian Brothers Neurosciences Institute Clinical Research, Elk Grove Village, Illinois
  - University of Kansas Alzheimer's Disease Center, Fairway, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - J. Gary Booker, MD APMC Clinical Drug Trials, Shreveport, Louisiana
  - Millennium Psychiatric Associates, Creve Coeur, Missouri
  - Atlantic Neuroscience Institute, Springfield, New Jersey
  - Neurological Associates of Albany, PC, Albany, New York
  - Parker Jewish Institute for Health Care and Rehabilitation, New Hyde Park, New York
  - Alzheimer's Memory Center, Charlotte, North Carolina
  - Neurobehavioral Clinical Research, Canton, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Sunstone Clinical Research, Medford, Oregon
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Neurology Clinic, PC, Cordova, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned: 250 subjects to be screened for a total of 140 subjects randomized 1:1:1 to one of three treatment arms: 20μg, 40μg or placebo Actual: 264 subjects were screened. 147 individual subjects were randomized and of those, 141 were dosed with trial drug.
Period: Overall Study
Arm/Group | Bryostatin 1 20ug | Bryostatin 1 40ug | Placebo
Started (Safety Analysis set) | 46 | 47 | 48
Completed | 38 | 29 | 39
Not Completed | 8 | 18 | 9
Not completed — Adverse Event | 2 | 4 | 5
Not completed — Withdrawal by Subject | 4 | 12 | 2
Not completed — noncompliance, investigator termination, | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bryostatin 1 20ug | Bryostatin 1 40ug | Placebo | Total
Number analyzed (Participants) | 46 | 47 | 48 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (8.40) | 70.2 (7.53) | 73.5 (7.68) | 71.7 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 23 | 71
  Male | 20 | 25 | 25 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 46 | 45 | 133
  African American | 3 | 1 | 3 | 7
  Asian | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 46 | 47 | 48 | 141
Mini Mental State Exam-version 2 (MMSE-2) baseline scores 4-9 [Count of Participants; unit: Participants] — ion, language, and praxis on a scale of 0-30. Lower scores indicate greater cognitive impairment. For this study, subjects were stratified at randomization based on Mini Mental State Exam version 2 (MMSE-2) scores 4-9 (severe cognitive impairment) and 10-15 (moderately severe impairment).
  Participants | 18 | 20 | 19 | 57
Mini Mental State Exam version 2 (MMSE-2) baseline score 10-15 [Count of Participants; unit: Participants] — For this study, subjects were stratified at randomization by Mini Mental State Exam version 2 (MMSE-2) scores 4-9 (severe cognitive impairment) and 10-15 (moderately severe impairment)
  Participants | 28 | 27 | 29 | 84

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Subjects With Treatment-emergent Adverse Events and Serious Adverse Events
Description: Evaluations of adverse events (AEs), serious adverse events (SAEs), Adverse event of special interest - myalgia
Time Frame: Baseline through 30 days post end of treatment (up to Day 107)
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Bryostatin 1 20ug | Bryostatin 1 40ug | Placebo
Number analyzed (Participants) | 46 | 47 | 48
participants
  Number of Subjects w Treatment Emergent AE (TEAE) | 30 | 39 | 28
  # of Subjects w Treatment Related TEAE | 17 | 24 | 8
  # of Subjects w TEAE leading to treatment discont. | 1 | 3 | 2
  # of Subjects with Serious TEAE | 1 | 6 | 3
  # of Subjects with Treatment Related Serious TEAE | 1 | 4 | 0
  # of Subjects w Treatment Emergent Myalgia | 1 | 4 | 0
  # of Subjects w Serious Treatment Emergent Myalgia | 0 | 0 | 0
  # of Subjects with Fatal TEAE | 0 | 1 | 0

2. Primary Outcome: Efficacy: Change From Baseline in Severe Impairment Battery (SIB) in the Full Analysis Set (FAS)
Description: The primary statistical objective for efficacy was to estimate the effect of bryostatin on the mean change in the total SIB score after 12 weeks of treatment, assessed at Week 13 (day 91). Efficacy analyses were conducted according to randomized groups. The SIB is used to assess cognition in subjects with moderate and severe AD. It is divided into nine subscales that include attention, language, orientation, memory, praxis, visuospatial ability, construction, social skills, orienting head to name. Non-verbal responses are allowed, thus decreasing the need for language output. Forty questions are included with a point score range of 0-100. Lower scores indicate greater cognitive impairment.
Time Frame: Primary analysis at Week 13 (day 91) after 12 weeks of treatment (up to day 107)
Population: The Full Analysis Set (FAS), consistent with a modified intention-to-treat principle (mITT), was defined as all randomized subjects who received at least one dose of randomized trial medication and who had at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: mean change from baseline in SIB score
Arm/Group | Bryostatin 1 20ug | Bryostatin 1 40ug | Placebo
Number analyzed (Participants) | 44 | 45 | 46
mean change from baseline in SIB score
  Week 13 Full Analysis Set (FAS): number analyzed (Participants) | 38 | 33 | 42
  Week 13 Full Analysis Set (FAS) | 1.6 (7.10) | 0.8 (6.58) | -0.4 (9.02)
  Week 13 Completer Analysis Set (CAS): number analyzed (Participants) | 38 | 33 | 42
  Week 13 Completer Analysis Set (CAS) | 1.6 (7.10) | 0.8 (6.58) | -0.7 (9.02)
  30-Day Followup Full Analysis Set: number analyzed (Participants) | 27 | 22 | 29
  30-Day Followup Full Analysis Set | 2.3 (8.17) | 0.6 (7.51) | -2.7 (11.44)
  30-Day Followup Completer Analysis Set: number analyzed (Participants) | 27 | 20 | 29
  30-Day Followup Completer Analysis Set | 2.3 (8.17) | 0.9 (7.85) | -2.7 (11.44)
Statistical Analysis 1: Comparison: Bryostatin 1 20ug vs Bryostatin 1 40ug vs Placebo; The primary statistical objective for efficacy was to estimate the effect of bryostatin on the mean change in the Severe Impairment Battery (SIB) after 12 weeks of treatment. A linear model was used for both estimation and significance testing. Primary analysis populations were defined as the Full Analysis Set (FAS) and the Completer Analysis Set (CAS); Test type: Superiority; p < 0.1, t-test, 1 sided — LSM and two-sided 80% CI were provided for treatment group differences and estimated endpoint values. A true mean difference in change from baseline in the SIB (one-sided at α=0.10) of at least 6.5 points in favor of bryostatin groups was assumed; Mean Difference (Net) = 6.5
Statistical Analysis 2: Comparison: Bryostatin 1 20ug vs Bryostatin 1 40ug vs Placebo; Change from baseline in SIB in the Completer Analysis Set (CAS); Test type: Superiority; p < 0.1, t-test, 1 sided; Mean Difference (Net) = 6.5

3. Secondary Outcome: Secondary Efficacy Endpoints
Description: * Change from baseline in the Severe Impairment Battery (SIB) at Weeks 5 and 9. Assesses cognition. Score range 0-100. Lower scores indicate greater cognitive impairment.
  * Change from baseline in Alzheimer Disease Cooperative Study Activities of Daily Living Inventory-Severe Impairment Version (ADCS-ADL-SEV) at Weeks 5, 9,13. A 19-item test of the performance of activities of daily living. Total score range 0-54; lower scores indicate greater functional impairment.
  * Change from baseline in MMSE-2 at Weeks 5, 9 and 13. Tests selected aspects of cognition on a scale of 0-30. Lower scores indicate greater cognitive impairment.
  * Change from baseline in Neuropsychiatric Inventory (NPI) at Weeks 5, 9,13. Caregiver interview assesses 12 behavioral disturbances. Scores range from 0-144; higher scores indicate greater behavioral disturbances.
  * Clinical Global Impression of Improvement (CGI-I) at Weeks 5, 9, 13. A 7-point scale range from (1) very much improved to (7) very much worse.
Time Frame: Week 5, Week 9, Week 13
Population: The number of participants analyzed over the course of the study diminished as a result of attrition.
Measure: Mean (Standard Deviation); unit: mean change from baseline
Arm/Group | Bryostatin 1 20ug | Bryostatin 1 40ug | Placebo
Number analyzed (Participants) | 46 | 47 | 48
mean change from baseline
  SIB Week 5 Full Analysis Set: number analyzed (Participants) | 44 | 44 | 46
  SIB Week 5 Full Analysis Set | 1.5 (7.36) | -0.8 (6.55) | -1.2 (10.31)
  SIB Week 5 Completer Analysis Set: number analyzed (Participants) | 38 | 32 | 42
  SIB Week 5 Completer Analysis Set | 1.7 (6.02) | 0.1 (5.93) | -1.9 (10.33)
  SIB Week 9 Full Analysis Set: number analyzed (Participants) | 38 | 38 | 43
  SIB Week 9 Full Analysis Set | 1.3 (6.87) | -0.2 (6.41) | -0.0 (9.91)
  SIB Week 9 Completer Analysis Set: number analyzed (Participants) | 37 | 33 | 42
  SIB Week 9 Completer Analysis Set | 1.2 (6.93) | -0.1 (6.06) | -0.1 (10.0)
  Week 5 ADCS-ADL-SIV : FAS: number analyzed (Participants) | 43 | 43 | 48
  Week 5 ADCS-ADL-SIV : FAS | -0.3 (4.16) | -1.1 (6.31) | -0.7 (5.07)
  Week 9 ADCS-ADL-SIV : FAS: number analyzed (Participants) | 37 | 38 | 43
  Week 9 ADCS-ADL-SIV : FAS | -1.4 (4.68) | -1.5 (5.05) | -1.3 (4.07)
  Week 13 ADCS-ADL-SIV : FAS: number analyzed (Participants) | 37 | 33 | 42
  Week 13 ADCS-ADL-SIV : FAS | -0.7 (4.59) | -1.0 (4.86) | -2.2 (5.28)
  Week 5 MMSE-2: FAS: number analyzed (Participants) | 44 | 44 | 46
  Week 5 MMSE-2: FAS | 0.4 (2.43) | -0.1 (2.79) | -0.1 (2.40)
  Week 9 MMSE-2: FAS: number analyzed (Participants) | 38 | 38 | 43
  Week 9 MMSE-2: FAS | 0.8 (2.98) | 0.3 (3.01) | 0.5 (3.11)
  Week 13 MMSE-2: FAS: number analyzed (Participants) | 38 | 33 | 42
  Week 13 MMSE-2: FAS | 0.5 (3.09) | 0.3 (2.54) | -0.2 (3.49)
  Week 5 Neuropsychiatric Inventory (NPI): FAS: number analyzed (Participants) | 41 | 41 | 44
  Week 5 Neuropsychiatric Inventory (NPI): FAS | -0.5 (11.72) | 1.7 (12.03) | -2.4 (10.31)
  Week 9 Neuropsychiatric Inventory (NPI): FAS: number analyzed (Participants) | 37 | 34 | 41
  Week 9 Neuropsychiatric Inventory (NPI): FAS | 0.5 (11.97) | 2.0 (8.33) | -2.5 (11.05)
  Week 13 Neuropsychiatric Inventory (NPI): FAS: number analyzed (Participants) | 37 | 32 | 39
  Week 13 Neuropsychiatric Inventory (NPI): FAS | 1.0 (12.62) | 2.0 (11.94) | 1.0 (10.45)

4. Post Hoc Outcome: Severe Impairment Battery (SIB) Scores by Memantine Use at Baseline
Description: Change from baseline in SIB score was compared between subjects receiving concurrent treatment with memantine and subjects not being treated with memantine.
Time Frame: Assessments at weeks 5, 9, 13, and 30 days after end of treatment (up to day 107).
Population: Participants in the 3 treatment groups were further sorted by use of memantine. The number of participants in each category at each timepoint is noted. Attrition occurred through the course of the study.
Measure: Mean (Standard Deviation); unit: mean change from baseline in SIB score
Groups:
- Bryostatin 1 20ug With Memantine: Bryostatin 20 micrograms administered IV over 45 minutes every other week after 2 initial loading doses of 24 micrograms administered weekly. A total of 7 doses administered over 12 weeks.
  Bryostatin 1: The investigational drug product, bryostatin, is a sterile, pyrogen-free, lyophilized powder intended for IV infusion upon reconstitution and dilution. Placebo is a sterile, pyrogen-free, lyophilized powder intended for IV infusion upon reconstitution and dilution.
- Bryostatin 1 40ug With Memantine: Bryostatin 40 micrograms administered IV over 45 minutes every other week after 2 initial loading doses of 48 micrograms administered weekly. A total of 7 doses administered over 12 weeks.
  Bryostatin 1: The investigational drug product, bryostatin, is a sterile, pyrogen-free, lyophilized powder intended for IV infusion upon reconstitution and dilution. Placebo is a sterile, pyrogen-free, lyophilized powder intended for IV infusion upon reconstitution and dilution.
- Placebo With Memantine: Placebo administered IV over 45 minutes every other week after 2 initial doses administered weekly. A total of 7 doses administered over 12 weeks.
  Placebo: The placebo is a sterile, pyrogen-free, lyophilized powder identical in appearance to the active drug, intended for IV infusion upon reconstitution and dilution.
- Bryostatin 1 20ug Without Memantine: Bryostatin 20 micrograms administered IV over 45 minutes every other week after 2 initial loading doses of 24 micrograms administered weekly. A total of 7 doses administered over 12 weeks.
- Bryostatin 1 40ug Without Memantine: Bryostatin 40 micrograms administered IV over 45 minutes every other week after 2 initial loading doses of 48 micrograms administered weekly. A total of 7 doses administered over 12 weeks.
- Placebo Without Memantine: Placebo administered IV over 45 minutes every other week after 2 initial doses administered weekly. A total of 7 doses administered over 12 weeks.
Arm/Group | Bryostatin 1 20ug With Memantine | Bryostatin 1 40ug With Memantine | Placebo With Memantine | Bryostatin 1 20ug Without Memantine | Bryostatin 1 40ug Without Memantine | Placebo Without Memantine
Number analyzed (Participants) | 26 | 37 | 31 | 18 | 8 | 15
mean change from baseline in SIB score
  Week 5 SIB change from Baseline: number analyzed (Participants) | 26 | 37 | 31 | 18 | 7 | 15
  Week 5 SIB change from Baseline | 0.1 (8.11) | -1.6 (6.50) | -1.3 (10.50) | 3.4 (5.75) | 3.9 (4.98) | -1.2 (10.26)
  Week 9 SIB change from Baseline: number analyzed (Participants) | 23 | 31 | 29 | 15 | 7 | 15
  Week 9 SIB change from Baseline | -0.1 (6.52) | -0.6 (6.88) | -0.4 (11.01) | 3.5 (7.04) | 2.0 (3.16) | 0.8 (7.44)
  Week 13 SIB change from Baseline: number analyzed (Participants) | 22 | 26 | 28 | 16 | 7 | 14
  Week 13 SIB change from Baseline | -0.5 (6.51) | -0.1 (6.61) | -0.5 (10.03) | 4.5 (7.01) | 3.9 (5.84) | -1.1 (6.89)
  30-day Followup SIB change from Baseline: number analyzed (Participants) | 15 | 20 | 18 | 12 | 2 | 11
  30-day Followup SIB change from Baseline | -1.1 (8.39) | 0.3 (7.71) | -3.8 (13.10) | 6.7 (5.58) | 4.0 (5.66) | -1.0 (8.31)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected beginning at the time of informed consent until the 30-day post treatment visit. For subjects enrolled under protocol versions 1 (17 Apr 2015) and 2 (20 Jan 2016), this collection occurred from Day -21 through Day 198 for subjects completing the study. For subjects enrolled under protocol version 3 (15 Jul 2016) this collection occurred from Day -28 through Day 105.
Description: In addition to the standard defined adverse events, an adverse event of special interest was defined in this study; myalgia.
Arm/Group | Bryostatin 1 20ug | Bryostatin 1 40ug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 1/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 2/46 | 6/47 | 4/48
Other Adverse Events (participants affected / at risk) | 21/46 | 46/47 | 12/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bryostatin 1 20ug (N=46) | Bryostatin 1 40ug (N=47) | Placebo (N=48)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Confusion postoperative (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dementia Alzheimer's Type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bryostatin 1 20ug (N=46) | Bryostatin 1 40ug (N=47) | Placebo (N=48)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (6) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 5 (5) | 1 (1)
Infusion site extravasation (General disorders) | 3 (3) | 3 (4) | 0 (0)
Fatigue (General disorders) | 1 (1) | 5 (5) | 0 (0)
Infusion site pain (General disorders) | 3 (3) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 4 (4)
Infusion site cellulitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (5) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 5 (5) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT02431468/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT02431468/SAP_001.pdf